CLINICAL TRIAL: NCT01596530
Title: A Randomised Double-Blind Placebo-controlled Multicentre Phase I Study to Assess the Biological Activity of AZD8931 in Patients With Early Breast Cancer Who Are Ineligible for Treatment With Trastuzumab as Defined by IHC Status
Brief Title: Evaluation of Drug Activity in Women With Breast Cancer and no Previous Herceptin Treatment
Acronym: CHIVE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: All AstraZeneca sponsored clinical trials of AZD8931 have been halted
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D0102C00019
Record Dates: First submitted 2012-04-27; First posted 2012-05-11 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Breast Neoplasm
Keywords: Breast Neoplasm; Breast Cancer; Breast Tumour; Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AZD8931 (Active Comparator): AZD8931
  Interventions: Drug: Drug-AZD8931
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Drug-Placebo

INTERVENTIONS:
Drug: Drug-AZD8931 — Active drug for biological activity
  Arms: AZD8931
Drug: Drug-Placebo — Placebo comparator for biological activity comparison
  Arms: Placebo

SUMMARY:
To compare the activity of AZD8931 against placebo on the cell markers in cancer tumours

DETAILED DESCRIPTION:
A Randomised Double-Blind Placebo-controlled Multicentre Phase I Study to Assess the Biological Activity of AZD8931 in Patients with Early Breast Cancer who are Ineligible for Treatment with trastuzumab as defined by IHC status

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 or older Early stage breast cancer and planned surgery
* Ineligible for Trastuzumab (Herceptin) treatment as per local guidelines
* World health Organisation performance status of 0 to 1 Tumour size amenable to obtaining adequate biopsies pre dosing.

Exclusion Criteria:

* Eligible for Trastuzumab (Herceptin) Treatment Known sensitivity to AZD8931, its excipients or drugs in its class;
* Including oral tyrosine kinase inhibitors History of eye conditions e.g. previous injury within 3 months or clinically significant eye disease
* Concurrent malignancy Unable to discontinue medication or herbal supplement known to inhibit CYP3A4 or CYP2D6

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effects of AZD8931 versus placebo on cytoplasmic p-MAPK after 7 days or more days of treatment | Day 7 - Day 14

SECONDARY OUTCOMES:
Comparison of the effects of AZD8931 versus placebo on p-EGFR, p-erbB2, p-erbB3 NUCLEAR p-Mapk, p-AKT and Ki67 after 7 or more days of treatment | Day 7 - Day 14
Assessment sof the safety and tolerability of AZD8931 as assessed by incidence of adverse events during the course of the study. | From study entry through to 30 days post treatment (Day 44 maximum)
Assessment of the plasma PK of AZD8931 | Day 1 - Day 14
Comparison of the effects of AZD8931 versus placebo on other biomarkers including but not limited to, erbB ligands, pER, PTEN, erbB receptor homo- and hetero- dimers, total MAPK, apoptosis markers and total AKT after 7 or more days of treatment. | Day 7 - Day 14
Establishing the baseline tumour characteristics, including but not limited to ER, PR and HER-2 status | Day -28 to Day 0
Exploration of the relationship between AZD8931 exposure (PK in plasma and tumour) and a selection of secondary biomarkers (e.g. p-EGFR, nuclear p-MAPK, Ki67 and apoptosis markers after ?7 days of treatment), if possible. | Day 1 - Day 14
Change from baseline in laboratory, vitals signs and ECG data | Day 1 - Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, M.D., Study Director — Internal
Locations (7):
- Germany (3):
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Wittenberg
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Yonsei
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei